CLINICAL TRIAL: NCT04800016
Title: Real-World Study of AcrySof™ IQ Vivity Extended Vision Intraocular Lenses (IOLs)
Brief Title: Real-World Study of Vivity Intraocular Lenses (IOLs)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Management decision. No patients enrolled
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILI875-P002
Record Dates: First submitted 2021-03-15; First posted 2021-03-16 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Aphakia; Presbyopia
Keywords: Cataract; Intraocular lens
MeSH Terms: conditions — Aphakia; Presbyopia; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Vivity IOL (Experimental): AcrySof IQ Vivity Extended Vision IOL implanted in the capsular bag in the posterior chamber of the eye during cataract surgery
  Interventions: Device: AcrySof IQ Vivity Extended Vision IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: AcrySof IQ Vivity Extended Vision IOL — UV and blue-light filtering extended depth of focus foldable IOL intended to provide a full range of vision from distance to functional near.
  Other Names: Model DFT015
Procedure: Cataract surgery — Cataract extraction by phacoemulsification, followed by implantation of the AcrySof IQ Vivity Extended Vision IOL

SUMMARY:
The primary objective of this clinical study is to assess the clinical performance of the AcrySof IQ Vivity Extended Vision IOL in a Chinese population.

DETAILED DESCRIPTION:
In this clinical study, subjects will be implanted with the AcrySof IQ Vivity Extended Vision IOL in both eyes. The second eye surgery will occur 7-28 days after the first eye. A total of 11 scheduled visits are planned, including a screening visit, two operative visits, and 8 postoperative visits. The total expected duration of the subject's participation will be about 13 months. This study will be conducted in China.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an approved informed consent;
* Willing and able to attend all scheduled study visits as required per protocol;
* Diagnosed with cataracts in both eyes;
* Pre-operative regular corneal astigmatism less than 1.0 diopter (D);
* Planned bilateral cataract removal by phacoemulsification.
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Glaucoma, diabetic retinopathy, retinitis pigmentosa and any pathologic changes associated with the optic nerve;
* Clinically significant corneal diseases;
* Clinically significant/severe dry eye that would affect study measurements based on the investigator's expert medical opinion;
* Previous intraocular surgery history;
* Pregnancy or lactation during study or planning to be pregnant/lactating;
* Systemic medications that, in the opinion of the Investigator, may confound the outcome or increase the risk to the subject;
* Other planned ocular surgical procedures;
* Patients who can only undergo cataract surgery in one eye.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Mean Monocular Distance Corrected Intermediate Visual Acuity (DCIVA) - First Eye | Month 6 post second eye implantation
  Intermediate visual acuity will be assessed at 66 centimeters (cm) with best correction of distance visual acuity in place. This endpoint is pre-specified for the first implanted eye.
Mean Monocular Distance Corrected Near Visual Acuity (DCNVA) - First Eye | Month 6 post second eye implantation
  Near visual acuity will be assessed at 40 centimeters (cm) with best correction of distance visual acuity in place. This endpoint is pre-specified for the first implanted eye.
  .
Incidence of ocular adverse events | Up to Month 12 post second eye implantation
  Ocular adverse events will be reported.
Incidence of secondary surgical interventions (SSIs) | Up to Month 12 post second eye implantation
  Secondary surgical interventions will be reported.
Incidence of severe or most bothersome visual disturbances (subjects surveyed with QUVID questionnaire) | Up to Month 12 post second eye implantation
  Subjects will be surveyed using the QUVID questionnaire.

SECONDARY OUTCOMES:
Percentage of Eyes Achieving 0.2 logMAR or better Best Corrected Distance Visual Acuity (BCDVA) - First Eye | Month 6 post second eye implantation
  Distance visual acuity will be assessed at 4 meters (m) with best correction of distance visual acuity in place. This endpoint is pre-specified for the first implanted eye.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Surgical, Study Director — Alcon (China) Ophthalmic Product Co., Ltd.
Locations (1):
- Hainan Bo'ao Super Hospital Co., Ltd., Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: No